CLINICAL TRIAL: NCT06488716
Title: A Phase Ia/Ib, Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Activity of RO7759065 as a Single Agent and in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of RO7759065 as a Single Agent and in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following a thorough review of safety data, preliminary efficacy data and an evaluation of overall risk-benefit, Sponsor made the decision to end the study.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO45296; 2024-513391-17-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-20; First posted 2024-07-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumour
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase Ia: Dose Escalation (Experimental)
  Interventions: Drug: RO7759065
- Phase Ia: Expansion (Experimental)
  Interventions: Drug: RO7759065
- Phase Ib: Dose Escalation (Experimental)
  Interventions: Drug: RO7759065; Drug: Atezolizumab
- Phase Ib: Expansion (Experimental)
  Interventions: Drug: RO7759065; Drug: Atezolizumab

INTERVENTIONS:
Drug: RO7759065 — Specified dose on specified days
Drug: Atezolizumab — Specified dose on specified days
  Arms: Phase Ib: Dose Escalation; Phase Ib: Expansion

SUMMARY:
This is a first-in-human Phase Ia/Ib, open-label, multicenter, dose escalation and dose expansion study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary anti-tumor activity of RO7759065 as a single agent (Phase Ia) or in combination with atezolizumab (Phase Ib) in patients with locally advanced, recurrent, or metastatic incurable solid tumor malignancies. Several key aspects of the study design and study population are summarized below.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end-organ function
* Measurable disease according to Response Evaluation criteria in Solid Tumors (RECIST) Version 1.1
* Histologically confirmed locally advanced, recurrent, or metastatic incurable solid tumor malignancy
* Availability of representative tumor specimens required for patients in select cohorts.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, and/or radiotherapy, within 3 weeks prior to initiation of study treatment
* Active hepatitis B or C or tuberculosis
* Positive test for human immunodeficiency virus (HIV) infection
* Acute or chronic active Epstein-Barr virus (EBV) infection at screening
* Administration of a live, attenuated vaccine (e.g., FluMist) within 4 weeks before first RO7759065 infusion
* Primary, untreated, or active central nervous system (CNS) metastases
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic stem cell or organ transplantation
* Any history of a Grade 3 immune-mediated adverse event attributed to prior cancer immunotherapy that resulted in permanent discontinuation of that agent
* Any history of a Grade 4 immune-mediated adverse event attributed to prior cancer immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants iwth Dose Limiting Toxicity (DLTs) | Up to approximately 5 years
Number of Participants with Adverse Events (AEs) | Up to approximately 5 years

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of RO7759065 | Up to approximately 5 years
Objective Response Rate (ORR) | Up to Approximately 5 Years
Duration of Response (DOR) | Up to approximately 5 years
Progression Free Survival (PFS) | Up to approximately 5 years
Percentage of Participants With Anti-Drug Antibodies (ADAs) to RO7759065 | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (11):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado, Aurora, Colorado
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Tennesse Oncology - NASH - SCRI - PPDS, Chattanooga, Tennessee
- St Vincent's Hospital Sydney, Darlinghurst, New South Wales, Australia
- Canada (3):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis Jewish General Hospital-3755 Cote Sainte-Catherine, Montreal, Quebec
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No